CLINICAL TRIAL: NCT00639509
Title: A Phase 2 Study of IMC-A12 (NSC742460) in Hepatocellular Carcinoma
Brief Title: IMC-A12 in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00283; NCI-2009-00283 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-08015; CDR0000589633; 08-015 (Other: Memorial Sloan-Kettering Cancer Center); 8124 (Other: CTEP); P30CA008748 (NIH); N01CM62206 (NIH)
Record Dates: First submitted 2008-03-19; First posted 2008-03-20 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cixutumumab

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Procedure: computed tomography; Procedure: contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
Procedure: computed tomography — Undergo contrast-enhanced computed tomography
  Other Names: tomography, computed
Procedure: contrast-enhanced magnetic resonance imaging — Undergo contrast-enhanced magnetic resonance imaging
  Other Names: Contrast-enhanced MRI

SUMMARY:
This phase II trial is studying how well IMC-A12 works in treating patients with advanced liver cancer. Monoclonal antibodies, such as IMC-A12, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (PFS) at 4 months in patients with advanced hepatocellular carcinoma (HCC) treated with anti-IGF-1R recombinant monoclonal antibody IMC-A12.

II. To determine the best overall response rate in patients treated with this drug.

SECONDARY OBJECTIVES:

I. To determine the median overall survival of patients treated with this drug. II. To evaluate the safety, tolerability, and adverse events profile of this drug in these patients.

III. To perform a subgroup analysis to compare PFS of patients with advanced HCC who are hepatitis B positive/hepatitis C negative versus patients who are hepatitis B negative/hepatitis C positive treated with this drug.

IV. To store pre-therapy paraffin embedded tumor tissue for future tissue-based correlative studies.

V. To evaluate tumor necrotic areas using a new volumetric method of assessing non-viable tumor as a correlate for response.

VI. To prospectively validate and compare the CLIP and the GDETCH staging systems and additional prognostic factors.

OUTLINE: Patients receive anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo serum sample collection at baseline for future tissue-based correlative studies. Previously collected paraffin embedded tumor tissue samples are also stored for future correlative studies.

After completion of study treatment, patients are followed every 3 months for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Unresectable, locally advanced, or metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Child's Pugh score A5, A6, B7, or B8
* No known brain metastases
* No history of primary CNS tumors
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 75,000/mcL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* PT/INR ≤ 1.7 times ULN
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Fasting serum glucose ≤ 125 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinical encephalopathy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-IGF-1R recombinant monoclonal antibody IMC-A12
* No poorly controlled diabetes mellitus

  * Patients with a history of diabetes mellitus are eligible provided their blood glucose is within normal range (fasting blood glucose < 120 mg/dL OR below ULN) and patient is on a stable dietary or therapeutic regimen for this condition
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* No history of seizures not well controlled with standard medical therapy
* No history of stroke
* No history of another primary cancer except for the following:

  * Curatively resected nonmelanoma skin cancer
  * Curatively treated carcinoma in situ of the cervix
  * Other primary solid tumor with no known active disease present that in the opinion of the investigator would not affect treatment outcome
* Prior local therapy (i.e., surgery, radiotherapy, hepatic arterial embolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) allowed provided the target lesion has not been treated with local therapy and/or the target lesion within the field of local therapy has shown an increase of ≥ 25% in size

  * At least 4 weeks since prior local therapy
* No prior systemic therapy except for sorafenib tosylate
* No prior agents targeting the IGF or IGF-1R pathway
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 03/06/2008 Primary Completion Date 02/08/2011 Recruitment Location is medical clinic
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Started | 24
Completed | 23
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- IMC-A12: Participants will receive IMC-A12 at a dose of 6mg/kg IV over 1 hour on Day 1 every week.
Arm/Group | IMC-A12
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.469631093)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: PFS Rate
Description: PFS defined as the time from first date of first treatment on the study until such time as progressive disease is confirmed or upon patient death if disease progression has not been evident at that time. A Simon's optimal two stage design will be used with the following assumption: a 4 months PFS of 62% is considered acceptable while a 4 months PFS of 42% is not acceptable.
Time Frame: At 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 23
percentage of participants | 30 [13 to 48]

2. Primary Outcome: Best Overall Response Rate (ORR)
Description: Best overall ORR will be defined as the proportion of patients achieving either confirmed partial response (PR) or confirmed complete response (CR). A Simon's optimal two stage design will be used with the following assumption: ORR of more than 20% is acceptable and an ORR less than 5% is not acceptable.
Time Frame: From the start of the treatment until disease progression/recurrence
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 23
participants | 0

3. Secondary Outcome: Median Overall Survival
Description: Median Overall Survival
Time Frame: Post-Treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 23
months | 8 [5.8 to 14]

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=24)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
ALT, SGPT (Investigations) | 3 (3)
AST, SGOT (Investigations) | 4 (4)
Alkaline Phosphatase (Investigations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Death not assoc w CTCAE term-Disease Progression (Gastrointestinal disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage, Rectum (Gastrointestinal disorders) | 1 (1)
Hemorrhage, Varices (esophageal) (Gastrointestinal disorders) | 1 (1)
Pain, Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelets (Investigations) | 1 (1)
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=24)
ALT, SGPT (Investigations) | 21 (21)
AST, SGOT (Investigations) | 23 (23)
Hypoalbuminemia (Metabolism and nutrition disorders) | 24 (24)
Alkaline phosphatase (Investigations) | 17 (17)
Hyperbilirubinemia (Investigations) | 21 (21)
Hypercholesterolemia (Investigations) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Investigations) | 9 (9)
Skin Disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Fatigue (General disorders) | 21 (21)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (24)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (17)
Hemorrhage (Blood and lymphatic system disorders) | 3 (3)
INR (Blood and lymphatic system disorders) | 15 (15)
Leukocyte count decrease (Investigations) | 10 (10)
Lymphocyte count decrease (Investigations) | 3 (3)
Serum Magnesium decrease (Metabolism and nutrition disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5)
Neurological disorder (Nervous system disorders) | 2 (2)
Neutrophil count decrease (Investigations) | 3 (3)
Activated partial thromboplastin prolonged time (Investigations) | 3 (3)
Pain-Abdomen NOS (Gastrointestinal disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Platelet count decrease (Investigations) | 19 (19)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 21 (21)
Vision blurred (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less